CLINICAL TRIAL: NCT03366792
Title: Comparative Analysis of Transperineal Versus Transrectal Approaches for MRI-Targeted Biopsy of the Prostate for the Detection and Characterization of Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigators chose to discontinue the study based on interim findings
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-01550
Record Dates: First submitted 2017-11-21; First posted 2017-12-08 (Actual); Results first posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MRI Targeted Biopsy (Experimental)
  Interventions: Device: Artemis™ software system

INTERVENTIONS:
Device: Artemis™ software system — Computerized targeting of mpMRI lesions. The computerized co-registration will then be performed by software within the Artemis™ system and will fuse the MR imaging with real-time ultrasound imaging.

SUMMARY:
The purpose of this study is to investigate a transperineal biopsy approach (outside of the rectum) using MRI targeting to facilitate better access to the whole prostate gland and provide limited risk of infectious complications after biopsy.

DETAILED DESCRIPTION:
Prostate cancer is the most common malignancy and the second most common cause of cancer death in men in the Western hemisphere. Definitive diagnosis of prostate cancer relies on biopsy of the prostate gland, which is historically performed by taking 12 random biopsies of the prostate by placing a needle through the rectum under ultrasound guidance. Recently, advances in MRI techniques have allowed identification of suspicious lesions within the prostate prior to biopsy, which has given rise to targeting biopsy cores to high-suspicion areas using fused ultrasound-MRI images. However, the most commonly used transrectal approach to biopsy is associated with a growing rate of infectious complications as well as poor sampling of the anterior region of the prostate, which is furthest from the rectum.

ELIGIBILITY:
Inclusion Criteria:

* No contraindication to prostate biopsy (e.g. coagulopathy, medical condition prohibiting abstinence from anti-platelet or anticoagulation therapies, anatomical considerations) Area of suspicion or known cancer focus on previously obtained mpMRI of the prostate (at least one lesion with MRI suspicion score >3/5)

Exclusion Criteria:

* Prior pelvic radiotherapy
* Evidence of urinary tract infection or significant urinary retention
* Prostate instrumentation (e.g. prostate biopsy, transurethral prostate procedure) within 2 months prior to mpMRI
* No evidence of suspicious lesions on mpMRI
* Irreversible coagulopathy
* Contraindication to sedation

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Taneja, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MRI Targeted Biopsy
Started | 46
Completed | 31
Not Completed | 15
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 2
Not completed — Ineligible (could not reach perinium) | 2
Not completed — Study Closure (interim analysis showed no significant results) | 4

BASELINE CHARACTERISTICS:
Arm/Group | MRI Targeted Biopsy
Number analyzed (Participants) | 31
Age, Continuous [Mean (Full Range); unit: years] | 66 [58 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Core Cancer Length
Description: Greater tumor length per core provides better diagnostic information. Data is reported as Transperineal (TP) core cancer length, Transrectal (TR) core cancer length, and for both (TP+TR)
Time Frame: 2 Months
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | MRI Targeted Biopsy
Number analyzed (Participants) | 31
mm
  TP | 5 [1.875 to 6.75]
  TR | 6 [2.1 to 7.75]
  TP+TR | 5 [1.95 to 7.25]

2. Secondary Outcome: Percentage of High-Grade Prostate Cancer Using Gleason Score
Description: High-grade prostate cancer is defined as a Gleason score > 6; a score that is the sum of the two Gleason grades assigned to a prostate tumor and that is based on a scale of 2 to 10 with the lowest numbers indicating a slow-growing tumor unlikely to spread and the highest numbers indicating an aggressive tumor.
  Data is reported as a percentage for Transperineal (TP), Transrectal (TR), and for both (TP+TR)
Time Frame: 2 Months
Measure: Number; unit: percentage of prostate cancer grades
Arm/Group | MRI Targeted Biopsy
Number analyzed (Participants) | 31
percentage of prostate cancer grades
  TP | 34
  TR | 40
  TP+TR | 49

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | MRI Targeted Biopsy
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 2/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MRI Targeted Biopsy (N=46)
Hematuria (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT03366792/Prot_SAP_000.pdf